CLINICAL TRIAL: NCT06609824
Title: Learn to Dare! Leiden
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University (Other)
Collaborators: Leids Universitair Behandel en Expertise Centrum (LUBEC) (Unknown)
Responsible Party: Principal Investigator, Anke M Klein, AS, Principal Inverstigator, Leiden University
Organization: Leiden University Medical Center (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2024-02-27-A.M. Klein-V2-5116
Record Dates: First submitted 2024-09-10; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Childhood Anxiety; Shyness
Keywords: Prevention; Childhood Anxiety; Shyness
MeSH Terms: conditions — Shyness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Group (Experimental): This arm consists of all participants who receive the training intervention. The purpose is to assess longitudinal effectiveness of the training within all participants.
  Interventions: Behavioral: Leer te Durven!

INTERVENTIONS:
Behavioral: Leer te Durven! — 'Leer te Durven!' is an eight-week preventative group training for children between the ages of 8 and 12. This training is evidence-based and is based on the principles of Cognitive Behavioral Therapy. With this program children learn to stand up for themselves in a safe environment, to face the situations that they find exciting and to be more confident in their own abilities. The training consists, among other things, of psychoeducation, exposure, and relaxation.

SUMMARY:
Research shows that many children face anxiety and stress related problems. However, as much as 70-80% of children do not receive help. The aim of this project is to offer a training for children who are hindered by their shyness or fears, so that all children can develop freely without being held back and so that the risk of escalation of fear and stress in the long term can be prevented. In this project the prevention training 'Learn to Dare!' will be offered to children between the ages of 8 and 18 where the long-term outcomes and the program itself will be evaluated for attractiveness and satisfaction. With the evidence-based program 'Learn to Dare!' children between the ages of 8 and 12 learn to stand up for themselves in a safe environment, to face the situations that they find exciting and to be more confident in their own abilities. This project aims to adapt the program so that it can be available up to and including 18 years in the future.

DETAILED DESCRIPTION:
Participants are recruited via the 'Knowledge Centre Anxiety and Stress in youth' (KAS) telephone line, by a research assistant or via the waiting list of LUBEC. Following recruitment, a research assistant conducts a screening call with the parent(s) lasting approximately half an hour to determine the child's eligibility for the project. Subsequently, the research assistant collaborates with a therapist from KAS/LUBEC to evaluate the case. If both agree that the child meets the criteria of the 'Learn to Dare!' program, the research assistant proceeds to conduct a diagnostic interview with both the child and parents. When the child still meets the requirements for 'Learn to Dare!', the therapist from LUBEC, who is going to give the trainings, will do an intake with the child and parents.

When the child still meets the criteria after this intake, a subsequent appointment will take place at LUBEC in Leiden, that serves as an opportunity for parents and children to familiarize themselves with the therapist and complete the baseline 1 measurement. This appointment will take about 1,5-2 hours. Two research assistants will administer questionnaires to the parent(s) and the child: demographics questionnaire, SCARED, CDI, WIRK-ALL. In addition, they will administer the anxiety scale of the SCID in combination with the ADIS severity index to the parent(s) and the child.

After baseline 1, there will be a waiting period of 4 weeks. After this period, the child and parents complete the SCARED questionnaire online (30 minutes) before commencing the treatment phase. The treatment comprises eight group sessions of 'Learn to Dare!' (one session per week; 1.5 hours each) along with assigned homework. After those eight weeks of treatment, the post-treatment session will take place at LUBEC (1,5-2 hours). The therapist will meet with the child and the parent(s) to evaluate the treatment together. The research assistants will administer the anxiety scale of the SCID in combination with the ADIS severity index to the parent(s) and the child. In addition, a couple of questionnaires will be administered: SCARED, CDI, WIRK-ALL, Training Evaluation Questionnaire. Lastly, there will be three follow-ups 6, 12, and 24 months after treatment (1,5 hours per follow-up). Parents have the option to conduct these follow-ups either at LUBEC or online. The anxiety scale of the SCID, along with the severity index of the ADIS questionnaire, is administered, along with supplementary questionnaires: SCARED, CDI, WIRK-ALL.

ELIGIBILITY:
Inclusion Criteria:

* Cut-off scores of the SCARED: for girls 31 and for boys 27.

Exclusion Criteria:

* Currently under treatment for anxiety complaints or under treatment in the mental health care system for other internalizing complaints.
* Anxiety problems or comorbid problems that require attention or treatment (including a 6 or higher on the severity index (CSR) of the ADIS and a score above the clinical cut-off on the Child Depression Inventory.)
* Difficulty in understanding the training.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety severity in children (SCARED-child) | During baseline 1, baseline 2, post-training, and the follow-ups (6, 12, and 24 months after the training)
  The Screen for Child Anxiety Related Disorders (SCARED) will be administered to the children. Scores on the SCARED range between 0-142. A higher score means higher anxiety levels.
Change in anxiety severity in children (SCARED-parent) | During baseline 1, baseline 2, post-training, and the follow-ups (6, 12, and 24 months after the training)
  The Screen for Child Anxiety Related Disorders (SCARED) will be administered to the parents. Scores on the SCARED range between 0-142. A higher score means higher anxiety levels.
Change in severity of anxiety in children (SCID-parent) | From baseline to the end of the training and follow-up (6, 12, and 24 months post-training).
  Severity of anxiety will be assessed using the Structured Clinical Interview for DSM Disorders (SCID) in combination with the severity index (Clinician Severity Rating) of the Anxiety Disorder Interview Schedule (ADIS-V). The CSR-score is a score between 0 and 8, with higher scores indicating a higher severity and interference of anxiety. The SCID will be administered to the parents.
Change in severity of anxiety in children (SCID-child) | From baseline to the end of the training and follow-up (6, 12, and 24 months post-training).
  Severity of anxiety will be assessed using the Structured Clinical Interview for DSM Disorders (SCID) in combination with the severity index (Clinician Severity Rating) of the Anxiety Disorder Interview Schedule (ADIS-V). The CSR-score is a score between 0 and 8, with higher scores indicating a higher severity and interference of anxiety. The SCID will be administered to the children.

SECONDARY OUTCOMES:
Change in self-efficacy of the children (WIRK-ALL child version) | From baseline to the end of the training and follow-up (6, 12, and 24 months post-training).
  The WIRK-all will be administered to the children to assess their change in self-efficacy. The WIRK-ALL is a short questionnaire and is an adaptation of the General Self-Efficacy Scale. The scores on the WIRK-ALL range between 10 and 40, with higher scores indicating higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Anke M Klein, AS, Principal Investigator — Leiden University
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
The investigators will share the data upon request, but only for specific purposes. In addition, the data needs to be deleted after use. The investigators will not share data that cannot be anonymised, such as the video data.

REFERENCES:
- [Background] Simon E, de Hullu E, Bogels S, Verboon P, Butler P, van Groeninge W, Slot W, Craske M, Whiteside S, van Lankveld J. Development of 'learn to dare!': An online assessment and intervention platform for anxious children. BMC Psychiatry. 2020 Feb 11;20(1):60. doi: 10.1186/s12888-020-2462-3. PMID 32046669